CLINICAL TRIAL: NCT03768232
Title: Ventilator Induced Diaphragm Dysfunction in Pediatric Critically Ill Patients
Brief Title: Ventilator Induced Diaphragm Dysfunction in Pediatric Critically Ill Patients (VIDD)
Acronym: VIDD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Matteo Di Nardo, Principal investigator, Bambino Gesù Hospital and Research Institute
Other Study IDs: 001
Record Dates: First submitted 2018-11-14; First posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Respiratory Failure; Respiratory Distress Syndrome; Mechanical Ventilation Complication
Keywords: ultrasound assessment; diaphragm disfuncion
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ultrasound asessment — US diaphragm measurements within 36 hours of initiation of MV. Measurements will be repeated daily for the duration of MV for the first week, then every 48 hours and 24 hours after the extubation.

SUMMARY:
evaluation of diaphragmatic disfunction eventually occurred in pediatric patient undergoing mechanical ventilation therapy

DETAILED DESCRIPTION:
Physician will perform US diaphragm measurements within 36 hours of initiation of MV. Measurements will be repeated daily for the duration of MV for the first week, then every 48 hours and 24 hours after the extubation.

Exposure to and duration of continuous NMBA infusion during the course of MV and use of CS will be recorded.

Ventilator logs and arterial gas analysis will be checked at the time of each US measurement to ascertain ventilator settings and SBF for the 24 hours preceding each US measurement.

Extubation success will be defined as no requirement for reintubation within 48 hours following extubation. The use of NIV immediately after extubation will be decided by the physician in charge according to the patient clinical history (presence of withdrawal syndrome, ect) and NOT according to DTF measurement.

ELIGIBILITY:
Inclusion Criteria:

* patients younger than 18 years old
* expected clinical requiring of invasive MV for more than 36 hours

Exclusion Criteria:

* neonates
* subjects with preexisting diagnoses of neuromuscular weakness
* diaphragm paresis
* chronic respiratory failure with ongoing requirement for invasive MV, or continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BiPAP) or with likely death within 48 hours.

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all patient admitted in PICU
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
measurement of occurrence rate of ventilator induced diaphragm disfunction in pediatric patient | through study completion an average of 100 days
  the assessment of the actual occurrence rate of VIDD in a population of PICU patients undergoing MV for acute respiratory failure of various etiology

SECONDARY OUTCOMES:
evaluation clinical impact of ventilator induced diaphragm disfunction in pediatric patient | through study completion an average of 100 days
  evaluation of the impact of VIDD and clinical outcomes of our patients in terms of Mechanical Ventilation free days
evaluation of two different diaphragmatic thickening fraction formula (DTF) | through study completion an average of 100 days
  evaluate the feasibility and clinical applicability of our formula for the calculation of DTF (mTdi-insp - mTdi-exp)/mTdi-med x 100, comparing it to the standard one (Tdi-insp - Tdi-exp)/Tdi-exp x 100.
evaluation clinical impact of ventilator induced diaphragm disfunction in pediatric patient | through study completion an average of 100 days
  evaluation of the impact of VIDD and clinical outcomes of our patients, in terms of MV free days, PICU length of stay (LOS) - days

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demoule A, Jung B, Prodanovic H, Molinari N, Chanques G, Coirault C, Matecki S, Duguet A, Similowski T, Jaber S. Diaphragm dysfunction on admission to the intensive care unit. Prevalence, risk factors, and prognostic impact-a prospective study. Am J Respir Crit Care Med. 2013 Jul 15;188(2):213-9. doi: 10.1164/rccm.201209-1668OC. PMID 23641946
- [Result] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Result] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Result] Francis CA, Hoffer JA, Reynolds S. Ultrasonographic Evaluation of Diaphragm Thickness During Mechanical Ventilation in Intensive Care Patients. Am J Crit Care. 2016 Jan;25(1):e1-8. doi: 10.4037/ajcc2016563. PMID 26724302
- [Result] Glau CL, Conlon TW, Himebauch AS, Yehya N, Weiss SL, Berg RA, Nishisaki A. Progressive Diaphragm Atrophy in Pediatric Acute Respiratory Failure. Pediatr Crit Care Med. 2018 May;19(5):406-411. doi: 10.1097/PCC.0000000000001485. PMID 29406380
- [Result] Goligher EC, Dres M, Fan E, Rubenfeld GD, Scales DC, Herridge MS, Vorona S, Sklar MC, Rittayamai N, Lanys A, Murray A, Brace D, Urrea C, Reid WD, Tomlinson G, Slutsky AS, Kavanagh BP, Brochard LJ, Ferguson ND. Mechanical Ventilation-induced Diaphragm Atrophy Strongly Impacts Clinical Outcomes. Am J Respir Crit Care Med. 2018 Jan 15;197(2):204-213. doi: 10.1164/rccm.201703-0536OC. PMID 28930478